CLINICAL TRIAL: NCT02213874
Title: The Influence of Trust in the Health Care System on Postpartum Contraceptive Choice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Angela Dempsey, Associate Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Dempsey-Trust Pro 12660
Record Dates: First submitted 2014-08-05; First posted 2014-08-12 (Estimated); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Contraception Behavior; Contraception
Keywords: Pregnant Women; Women's Health; Contraception; Trust in Health Care
MeSH Terms: conditions — Contraception Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Questionnaire (Other): A questionnaire will be administered during the early stages of prenatal care & again during the postpartum period. The initial questionnaire will assess trust in the health care system, locus of control, religiosity, health literacy & collect information about demographics, contraceptive & reproductive history, future pregnancy intentions, & baseline knowledge about contraception. The postpartum questionnaire will repeat questions about future pregnancy & contraception intentions, trust in the health care system, knowledge of contraception and collect new information about characteristics of antenatal contraceptive counseling received including whether a provider recommended a specific method of contraception, the amount of counseling received, & the type of counseling received.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire will be administered during the early stages of prenatal care & again during the postpartum period. The initial questionnaire will assess trust in the health care system, locus of control, religiosity, health literacy & collect information about demographics, contraceptive & reproductive history, future pregnancy intentions, & baseline knowledge about contraception. The postpartum questionnaire will repeat questions about future pregnancy & contraception intentions, trust in the health care system, knowledge of contraception and collect new information about characteristics of antenatal contraceptive counseling received including whether a provider recommended a specific method of contraception, the amount of counseling received, & the type of counseling received.

SUMMARY:
The purpose of this research is to understand the relationship between trust in the health care system and choice of contraception during the postpartum period among pregnant women receiving prenatal care.

Research subjects will complete a questionnaire at enrollment and between delivery and within 5 days of hospital discharge.

A chart review will also be completed to gather use of a birth control method at the six week postpartum visit as well as pertinent medical diagnoses and recorded data such as height, weight, body mass index, and contraceptive plan as documented in the postpartum medical chart.

DETAILED DESCRIPTION:
The aims of the proposed research are three-fold:

1. To identify whether trust in the health care system is associated with choice of the highest efficacy contraception (intrauterine contraception, implantable contraception, and sterilization) in the immediate postpartum period among pregnant women receiving prenatal care.
2. To explore which patient-level factors (sociodemographic, reproductive history, future pregnancy intentions) and provider-level factors (antenatal contraceptive counseling) are associated with choice of the highest efficacy contraception in the immediate postpartum period among pregnant women receiving prenatal care.
3. To determine whether trust in the health care system is altered during the receipt of prenatal care or delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women receiving prenatal care at Medical University of South Carolina (MUSC)
* Age 18 or older

Exclusion Criteria:

* Greater than 20 weeks gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Choice of long acting contraception (IUD or implant) for postpartum contraception | immediately postpartum
  Using a questionnaire adminstered immediately postpartum, we will ascertain whether participants indicate plan to use either an IUD or implant for contraception. We will also measure use of IUD or implant through chart abstraction of their 6 week postpartum visit.

SECONDARY OUTCOMES:
Trust in the health care system | immediately postpartum
  We will also evaluate trust as an outcome and evaluate whether certain patient-level or antepartum care characteristics predict higher levels of trust. Trust is measured through a validated scale containing 17 questions measured using a likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Angela Dempsey, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC Women's Health, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No